CLINICAL TRIAL: NCT02928991
Title: Fludarabine-Based Conditioning for Matched Related Donor Bone Marrow Transplantation in Patients With Bone Marrow Failure Syndromes
Brief Title: Fludarabine Based RIC for Bone Marrow Failure Syndromes
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Principal Investigator, Timothy Olson, Assistant Professor, Children's Hospital of Philadelphia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-011465; 14BT057 (Other: Children's Hospital of Philadelphia)
Record Dates: First submitted 2016-10-07; First posted 2016-10-10 (Estimated); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Bone Marrow Failure Syndromes
Keywords: Acquired aplastic anemia; Inherited bone marrow failure
MeSH Terms: conditions — Bone Marrow Failure Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (3):
- Acquired Aplastic Anemia (AA) (Experimental): Patients with severe or very severe acquired aplastic anemia (AA). Patients will receive a matched related donor bone marrow transplant following reduced intensity conditioning (RIC) including thymoglobulin (ATG), fludarabine and dose-reduced cyclophosphamide.
  Interventions: Other: MRD-BMT with Fludarabine-based RIC for Acquired AA
- Inherited Bone Marrow Failure Syndrome + Trilineage Aplasia (Experimental): Patients with inherited bone marrow failure (iBMF) syndromes with trilineage aplasia includes those with diagnoses of Fanconi Anemia, Dyskeratosis Congenita, and related conditions. Patients will receive a matched related donor bone marrow transplant following conditioning with fludarabine, cyclophosphamide, thymoglobulin.
  Interventions: Other: MRD-BMT with Fludarabine-based RIC for iBMF with trilineage aplasia
- Inherited Bone Marrow Failure Syndrome no Trilineage Aplasia (Experimental): Patients with inherited bone marrow failure (iBMF) syndromes without trilineage aplasia includes those with diagnoses of Severe Congenital Neutropenia, Diamond-Blackfan Anemia, and related conditions. Patients will receive a matched related donor bone marrow transplant following conditioning with thymoglobulin, busulfan and fludarabine.
  Interventions: Other: MRD-BMT with Fludarabine-based RIC for iBMF without trilineage aplasia

INTERVENTIONS:
Other: MRD-BMT with Fludarabine-based RIC for Acquired AA — Fludarabine: Dose: 30mg/m2/day (<10kg will receive 1mg/kg/day) Days: -7, -6, -5, -4, -3
  Cyclophosphamide: Dose: 60mg/kg/day Days: -5, -4
  Thymoglobulin: Dose: 3mg/kg/day Days: -4, -3, -2
  Bone marrow infusion: Day 0
  Arms: Acquired Aplastic Anemia (AA)
Other: MRD-BMT with Fludarabine-based RIC for iBMF with trilineage aplasia — Fludarabine: Dose: 30mg/m2/day (<10kg will receive 1mg/kg/day) Days: -7, -6, -5, -4, -3
  Cyclophosphamide: Dose: 10 mg/kg/day Days: -6, -5, -4, -3
  Thymoglobulin: Dose: 3mg/kg/day Days: -4, -3, -2
  Bone marrow infusion: Day 0
  Arms: Inherited Bone Marrow Failure Syndrome + Trilineage Aplasia
Other: MRD-BMT with Fludarabine-based RIC for iBMF without trilineage aplasia — Fludarabine: Dose: 30mg/m2/day (<10kg will receive 1mg/kg/day) Days: -6, -5, -4, -3, -2
  Busulfan: Dose: every 6 hours for a total of 12 doses with dosing adjustments to achieve a steady state concentration of 900-1200ng/mL OR daily for a total of 3 doses targeting AUC 3600-6000 (micromole/liter)*minute Days: -7, -6, -5, -4
  Thymoglobulin: Dose: 3mg/kg/day Days: -10, -9, -8
  Bone marrow infusion: Day 0
  Arms: Inherited Bone Marrow Failure Syndrome no Trilineage Aplasia

SUMMARY:
This is a pilot study to determine whether fludarabine-based reduced intensity conditioning (RIC) regimens facilitate successful donor engraftment of patients with acquired aplastic anemia (AA) and Inherited bone marrow failure (iBMF) syndromes undergoing Matched related donor bone marrow transplant (MRD-BMT).

DETAILED DESCRIPTION:
Acquired AA patients will receive the experimental regimen of fludarabine with dose-reduced cyclophosphamide, with results in this prospective single arm experimental group evaluated in the context of our institutional historical experience using HD Cy regimens as well as published outcomes using both fludarabine and high-dose cyclophosphamide-based regimens for MRD-BMT in aplastic anemia. iBMF syndrome patients will receive one of two fludarabine-containing regimens based on disease characteristics, and our outcomes will be compared to previously published data using a variety of regimens. Graft versus host disease (GvHD) prophylaxis will consist of cyclosporine/tacrolimus alone for patients with acquired AA or cyclosporine/tacrolimus plus mycophenolate for patients with iBMF syndromes. For both acquired AA and iBMF syndrome patients, donor chimerism will be assessed at scheduled intervals following BMT and will be used to define patients with full donor or mixed chimerism for comparisons of survival, graft failure, cytogenetic, GvHD, and immune reconstitution outcomes.

ELIGIBILITY:
Patients 0-22 years with acquired aplastic anemia or a diagnosed inherited bone marrow failure syndrome, and a fully Human leukocyte antigen (HLA)-matched (10/10) related donor.

Inclusion Criteria:

Patient:

1. Ages 0-22 years at time of enrollment
2. Diseases:

   * Patients with severe or very severe acquired AA, defined by:

     * Bone marrow biopsy demonstrating cellularity of <25% (at least 2 weeks from last dose of G-CSF), in addition to 2 of the following: absolute neutrophil count (ANC) <500/µL, platelets < 20,000/µL and absolute reticulocytes <40,000/µL
     * Negative evaluation for inherited bone marrow failure conditions and negative evaluation for dysplasia or cytogenetic abnormalities associated with myelodysplastic syndromes
     * Patients with concurrent paroxysmal nocturnal hemoglobinuria (PNH) clones are eligible, as long as they meet criteria for severe or very severe aplastic anemia as defined above
   * Patients with clinically diagnosed and/or genetically proven iBMF syndromes, resulting in chronic red blood cell or platelet-transfusion dependence and/or an absolute neutrophil count <500/µL. These disorders include, but are not limited to:

     * Fanconi Anemia
     * Dyskeratosis Congenita
     * Severe Congenital Neutropenia
     * Diamond-Blackfan Anemia
     * Congenital Dyserythropoietic/Sideroblastic Anemias
     * Congenital Amegakaryocytic Thrombocytopenia
     * Shwachman-Diamond Syndrome
3. Lansky or Karnofsky performance >60
4. HLA matched related donor available.
5. No active untreated infection
6. Females of childbearing potential must have negative pregnancy test.

Organ Function:

* Serum creatinine <1.5xupper limit of normal for age Hepatic: Transaminases <5x normal
* Cardiac shortening fraction >27%
* Bilirubin <2.5x normal (unless elevation due to Gilberts disease).

Donor Selection Criteria:

* Donor selection will comply with U.S. Food and Drug Administration's Code of Federal Regulations
* Fully HLA-matched related donor.
* Donor must be at least 6 months of age
* Donor suitable for bone marrow collection and meets eligibility for donation, including fulfilling infectious disease criteria as per SOP, including HIV, Hepatitis B, Hepatitis C Polymerase chain reaction (PCR) negative.
* If subject has confirmed iBMF syndrome, donor must be evaluated for this disorder and testing must be negative
* Children's Hospital of Philadelphia (CHOP) bone marrow transplant (BMT) procedures apply for determining donor eligibility, including donor screening and testing for relevant communicable disease agents and diseases.
* Donor evaluation and collection procedure as per CHOP Standard Operating Procedures (SOP)

Exclusion Criteria:

* Uncontrolled bacterial, viral or fungal infections
* HLA matched related donor unable to donate bone marrow.
* No eligible fully HLA-matched related donor
* Pregnant females
* Patients with a clinical diagnosis of Myelodysplastic syndrome (MDS) defined by combination of bone marrow dysplasia and classic cytogenetic lesion (Monosomy 7, Trisomy 8 eg.), with or without excess blasts.
* Patients with PNH without underlying bone marrow aplasia

Max Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Estimated)
Dates: Start 2015-04; Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Rate of graft failure | Up to 1 year post transplant
  Combined rate of primary and secondary graft failure. Primary graft failure is defined as no evidence of neutrophil engraftment by day +28 after stem cell infusion. Secondary graft failure is defined as an ANC<100 for >7-10 days after initial engraftment occurs and is confirmed by hypocellular bone marrow biopsy and donor engraftment <20%.
Time to neutrophil engraftment | Up to 1 year post transplant
  The time from the day of transplant until neutrophil engraftment, which is defined as the first day of ANC >500/ul for the first of 3 consecutive days.
Transplant-related mortality | Up to 100 days post transplant

SECONDARY OUTCOMES:
Rate of overall survival | Up to 1 year post transplant
Rate of disease free survival | Up to 1 year post transplant

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Olson, MD, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No